CLINICAL TRIAL: NCT00152347
Title: A Double-Blind, Randomized Control Trial Comparing Botulinum Toxin Type A (Botox) and Placebo in the Treatment of Idiopathic Clubfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H05-70384
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Idiopathic Clubfoot (Talipes Equinovarus)
MeSH Terms: conditions — Clubfoot | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botox — See Detailed Description

SUMMARY:
The purpose of this study is to continue the work from the previous review study and determine the effectiveness of Botox in treating patients with idiopathic clubfoot by comparing outcomes of subjects treated with manipulation and casting plus Botox (treatment group) to those treated with manipulation and casting plus placebo (control group).

The null hypothesis is that manipulation and casting plus Botox is not an effective treatment for idiopathic clubfoot. The alternate hypothesis is that manipulation and casting plus Botox is an effective treatment for idiopathic clubfoot.

DETAILED DESCRIPTION:
The study timeline is divided into five phases which have been defined based on experiences with the previous review and with clubfoot treatment in general. These phases are as follows: 1) study treatment (Botox injection versus placebo); 2) post-treatment manipulation and casting; 3) bracing and full-time maintenance; 4) intent-to-treat intervention for management of first-time non-responders (NR1) and first-time recurrences (Rec1) post-study treatment; and 5) rescue intervention for management of second-time non-responders (NR2) and second-time recurrences (Rec2) post intent-to-treat intervention.

We will utilize a double-blind randomized control trial to assess the efficacy of Botox in the treatment of idiopathic clubfoot. Patients, parents, both participating surgeons, and members of their clinical and research teams (physiotherapist, occupational therapist, orthopaedic technologist, orthotist, research assistant) will be blinded to the study group (Botox group versus control group) each subject belongs in. The pharmacist preparing the syringes for injection will not be blinded.

Subjects will be randomly assigned to receive either Botox (Treatment group) or placebo injection (Control group). Subjects in the treatment group will receive Botox injections dosed at 10 IU/kg prepared by diluting 100 IU of Botox in 1cc of unpreserved saline. If the child has bilateral clubfoot, the contents will be divided equally for injection into each gastrocnemius. Placebo injections for the control group will contain unpreserved saline at 0.1cc/kg (such that a 4.5 kg subject will receive 0.45cc).

ELIGIBILITY:
Inclusion Criteria:

1. children presenting with idiopathic clubfoot at BC Children's Hospital and Hospital for Sick Children
2. children ranging in age from 1 day to 2 months old
3. children who have reached hindfoot stall
4. children with complete pre-study data *From protocol, hindfoot stall is defined: "following initial manipulation and casting of clubfoot, when the forefoot can be abducted beyond 60 degrees but hindfoot equinus persists, requiring need for further intervention to correct the clubfoot deformity"

Exclusion Criteria:

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2005-09; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Response to study treatment (as indicated by ankle dorsiflexion with knee in flexion of 15 degrees or greater)

SECONDARY OUTCOMES:
Patient outcomes collected at every patient visit including:
1. Ankle dorsiflexion with knee in extension
2. Plantarflexion
3. Heel bisector scores
4. Occurrence of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, FRCSC, MSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada